CLINICAL TRIAL: NCT06164925
Title: Standardising and Simplifying the Global Leadership Initiative on Malnutrition (GLIM) for Its More General Application
Status: Recruiting | Type: Observational
Sponsor: University of Tartu (Other)
Collaborators: Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Alastair Forbes, Visiting Professor, University of Tartu
Other Study IDs: 23092
Record Dates: First submitted 2023-11-01; First posted 2023-12-11 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-02

CONDITIONS: Malnutrition
Keywords: GLIM criteria; GLIM; nutrition assessment; nutrition screening; muscle mass
MeSH Terms: conditions — Malnutrition | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Inpatients of the Tartu University Hospital: Inclusion Criteria:
  Age of 18+ years, able and willing to sign the consent form, inpatients of the Tartu University Hospital, admitted within 72 hours before enrolment.
  Exclusion Criteria:
  Age of <18 years, inability or refusal to sign the consent form, pregnant or lactating women, more than 72 hours passed since admission, patients isolating with an infection.
  Interventions: Diagnostic Test: Nutrition screening and assessment

INTERVENTIONS:
Diagnostic Test: Nutrition screening and assessment — The patient is interviewed for changes in body weight in the last six months and food intake in the last two weeks.
  The investigator evaluates the patient's diet, symptoms related to their nutritional status, and functional capacity according to the Subjective Global Assessment (SGA). The SGA tool itself is completed by the researcher.
  Height and weight of the patient are measured, if not yet recorded, and BMI is calculated.
  The patient's muscle mass is measured using mid-upper arm circumference (MUAC), calf circumference (CC) and bioelectrical impedance (BIA), and their muscle function assessed using hand grip strength.

SUMMARY:
This observational study of aims to test whether and how the results of GLIM change when using different approaches and methods to carry out its components.

DETAILED DESCRIPTION:
The main questions the study aims to answer are:

* What is the most effective pre-GLIM screening approach?
* Which of the simple, globally accessible muscle mass measurement methods works the best in the context of GLIM?
* How does using simpler approaches to screening and muscle mass measurement affect the performance of GLIM in detecting Subjective Global Assessment (SGA) defined malnutrition and 1-year mortality?

Participants will be/have:

* asked questions about their recent food intake and possible non-volitional weight loss
* assessed for malnutrition with SGA
* weighed, and their height will be measured (if not already recorded)
* their muscle mass measured with a measuring tape (mid-upper arm circumference and calf circumference) and bioelectrical impedance
* their muscle function measured using hand grip strength
* have their patient records looked at to extract their weight and height data (if present), diagnoses, routine blood test results, abdominal computed tomography (CT) scan (if present), dual-energy x-ray absorptiometry (DEXA) scan (if present), 1-year mortality and personal identification code for documentation (the latter will be deleted when the study period is over).

ELIGIBILITY:
Inclusion Criteria:

* Age of 18+ years
* Able and willing to sign the consent form
* Inpatients of the Tartu University Hospital
* Admitted within 72 hours before enrolment

Exclusion Criteria:

* Age of <18 years
* Inability or refusal to sign the consent form
* Pregnant or lactating women
* More than 72 hours passed since admission
* Patients isolating with an infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients of day patients admitted to the Tartu University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Subjective Global Assessment (SGA) defined malnutrition | baseline, pre-intervention/procedure/surgery
  Subjective Global Assessment (SGA) can be considered a method that is close to a "gold standard" for malnutrition assessment. Therefore, the study will analyse how different approaches to screening and muscle mass measurement affect the performance of GLIM in detecting Subjective Global Assessment (SGA) defined malnutrition.
One-year mortality | through study completion, an average of 1 year
  One year after the data collection, we will look at the patient records to collect the 1-year mortality data. This will give information about whether and how different approaches to components of GLIM affect its ability to predict one-year mortality.
Computed tomography (CT) defined muscle mass | baseline, pre-intervention/procedure/surgery
  One of the GLIM criteria is "reduced muscle mass", and this study will investigate how muscle mass measured with simpler methods compares against muscle mass measured with CT.
DEXA defined muscle mass | baseline, pre-intervention/procedure/surgery
  One of the GLIM criteria is "reduced muscle mass", and this study will investigate how muscle mass measured with simpler methods compares against muscle mass measured with DEXA.

SECONDARY OUTCOMES:
Bioelectrical impedance (BIA) defined muscle mass | baseline, pre-intervention/procedure/surgery
  One of the GLIM criteria is "reduced muscle mass", and this study will investigate how muscle mass measured with simpler methods compares against muscle mass measured with BIA.

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Forbes, MD, Principal Investigator — University of Tartu, Tartu University Hospital
Locations (1):
- Tartu Ülikooli Kliinikum, Tartu, Tartu, Estonia